CLINICAL TRIAL: NCT03528798
Title: Analysis of Medication Data With the ApoMining-Database - - A Retrospective Analysis of Data From BioCog Study
Brief Title: Analysis of Medication Data With the ApoMining-Database
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine Berlin (CCM, CVK), Charite University, Berlin, Germany
Other Study IDs: ApoMining
Record Dates: First submitted 2018-04-24; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to analyse medication data from the BioCog Study with the ApoMining-Database and to determine the positive and negative predictive value from the ApoMining-Database for prediction of postoperative delirium (POD).

DETAILED DESCRIPTION:
From 2014-2017 the BioCog Study (ClinicalTrials.gov Identifier: NCT02265263) collected data from 439 perioperative elderly patients in Campus Virchow - Klinikum, Universitätsmedizin Berlin. According to the study protocol, a delirium assessment was performed each day after operation until the 7th postoperative day. At this time, it is known which patients developed postoperative delirium (POD) and which did not. Additionally, from each patient data on long-term medication before operation and applied medication during operation and in the recovery room were collected. In this study, the investiagtors analyse the long-term medication and the perioperative medication from BioCog-Study patients with the ApoMining-Database (http://www.apothesen.de/index.php?id=878; ApoThesenGmbH; Bad Münstereifel; Germany). The ApoMining-Database is a medication database, which analyse tolerability and risks of medications for the elderly. The database generates a hit once a medication reveal a risk for delirium. Additionally, the database can calculate the anticholinergic burden of the medication according to the prescribing information. Whereas the investigators already know, which patient developed a POD, they will determine positive and negative predictive value from the ApoMining-Database for prediction of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* From BioCog study (NCT02265263)

Exclusion Criteria:

* From BioCog study (NCT02265263)

Additionally for this analysis:

Inclusion criteria:

• Enrollment at Campus Virchow - Klinikum, Charité - Universitätsmedizin Berlin

Exclusion criteria:

* No delirium assessment
* No long-term medication before operation

Ages: 65 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing elective surgery
Sampling Method: Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of postoperative delirium | Up to 7 days after surgery
  Positive predictive value of the application of the ApoMining-Database for prediction of postoperative Delirium (the prediction of delirium by Apomining data base compared to occurence of Delirium in BioCog study)

SECONDARY OUTCOMES:
Negative predictive value of postoperative delirium | Up to 7 days after surgery
  Negative predictive value of the application of the ApoMining-Database for prediction of postoperative delirium.
Cholinesterase activity | Before surgery, one day after surgery, 3 months after surgery
  Cholinesterase activity is assessed by Acetylcholinesterase and Butyrylcholinesterase within the BioCog study
Delirium | Up to 7 days after surgery
  Delirium is defined within the BioCog study: according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) and/or as ≥ 2 cumulative points in the nursing Delirium Screening Scale (Nu-DESC) and/or a positive Confusion Assessment Method (CAM) and/or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score and/or patient chart review that shows descriptions of delirium.

OTHER OUTCOMES:
Anticholinergic burden | One day before surgery
  Anticholinergic burden is calculated by the ApoMining-Database
Delirium prediction | Up to the end of stay in the recovery room, an expected average of 1 day
  Delirium prediction is calculated by Apomining database.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite - Universitätsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine Berlin (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No